CLINICAL TRIAL: NCT02982018
Title: Clinical Evaluation of Approved and Investigational Contact Lenses Using New UV Additive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5638
Record Dates: First submitted 2016-10-31; First posted 2016-12-05 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Investigational Contact Lens with UV Blocker (Experimental): Subjects will be dispensed the investigational contact lens with UV blocker to wear daily for a period of 12 weeks with follow-up visits occurring after 1, 2, 4, 8, and 12 weeks. Afterwards, the subjects will wear their habitual contact lenses for a period of two weeks with weekly visits.
  Interventions: Device: senofilcon A with new UV blocker
- Marketed Contact Lens (Active Comparator): Subjects will be dispensed the marketed contact lens to wear daily for a period of 12 weeks with follow-up visits occurring after 1, 2, 4, 8, and 12 weeks. Afterwards, the subjects will wear their habitual contact lenses for a period of two weeks with weekly visits.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A with new UV blocker — Investigational Contact Lens
  Arms: Investigational Contact Lens with UV Blocker
Device: senofilcon A — J&J Marketed Contact Lens
  Arms: Marketed Contact Lens

SUMMARY:
Randomized, 8-visit dispensing study over 14 weeks to evaluate the safety and efficacy of an investigational contact lens with a new UV blocker compared to a marketed contact lens.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read and sign the Informed Consent form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Healthy adult males or females age ≥ 18 years of age with signed informed consent. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them.
4. The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and - 6.00 Diopters (D).
5. The subject's refractive cylinder must be ≤ 1.00 D in each eye.
6. The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
7. Subjects should own a wearable pair of spectacles.
8. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of Daily Wear per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis.
9. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week.
10. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g. Seldane, Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication.
4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
5. Any previous, or planned, ocular or interocular surgery (e.g.., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.).
6. Any grade 2 or greater slit lamp findings (e.g.., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g.., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
7. Any known hypersensitivity or allergic reaction to Optifree®Puremoist® multi-purpose care solution or Eye-Cept® rewetting drop solution.
8. Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
9. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
10. Toric, extended wear, monovision or multi-focal contact lens correction.
11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
12. History of binocular vision abnormality or strabismus.
13. Employee or relative of employees of sponsor or investigational clinic (e.g., Investigator, Coordinator, Technician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-02-18 (Actual); Study Completion 2017-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Jacksonville, Florida
  - Longwood, Florida
  - Sarasota, Florida
  - Closter, New Jersey
  - Vestal, New York
  - Pickens, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 133 subjects were enrolled into the study. Of the enrolled subjects 131 were dispensed study lenses and 2 subjects failed to meet the eligibility criteria. Of the dispensed subjects 123 completed the study and 8 subjects were discontinued.
Groups:
- Senofilcon A With New UV Blocker: Subjects that wore the senofilcon A with new UV blocker lens throughout the entire duration of the study.
- Senofilcon A: Subjects that wore the senofilcon A lens throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Senofilcon A With New UV Blocker | Senofilcon A
Started | 67 | 64
Completed | 62 | 61
Not Completed | 5 | 3
Not completed — Incorrect Lens Dispensed | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lens Discomfort | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon A With New UV Blocker | Senofilcon A | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.2 (8.15) | 32.1 (7.99) | 31.6 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 47 | 92
  Male | 22 | 17 | 39
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 6 | 1 | 7
  Black or African American | 4 | 1 | 5
  White | 56 | 62 | 118
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Eyestrain Related to Glare
Description: Eyestrain related to glare was assessed at the 2-, 4-, 8- and 12- week follow-up visits using an 11-item questionnaire. This questionnaire assesses patient-experience attributes of soft contact lenses. Derived eyestrain related to glare scores using Item Response Theory (IRT) follow a normal distribution with a mean of 50 and a standard deviation of 10. Scores in this study ranged from 30 to 70. Lower scores indicate better performance. This questionnaire is still under development and the data collected is considered exploratory.
Time Frame: Up to 12-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Senofilcon A With New UV Blocker (Test): Subjects that wore the senofilcon A with new UV blocker lens for the first 12-weeks of the study.
- Senofilcon A (Control): Subjects that wore the senofilcon A lens for the first 12 weeks of the study.
Arm/Group | Senofilcon A With New UV Blocker (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 61 | 59
Units on a Scale
  2-Week Follow-up | 44.64 (6.562) | 45.37 (7.631)
  4-Week Follow-up | 46.40 (7.489) | 44.59 (7.300)
  8-Week Follow-up | 44.67 (6.751) | 43.57 (6.012)
  12-Week Follow-up | 43.66 (5.921) | 44.02 (7.687)

2. Primary Outcome: Distance Monocular logMAR Visual Acuity (VA)
Description: Distance logMAR Visual Acuity was assessed for each subject and eye at 2-, 4- 8- and 12-weeks. The average logMAR visual acuity for each lens and time point was reported. Lower values of logMAR indicate better vision.
Time Frame: Up to 12-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Senofilcon A With New UV Blocker (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 61 | 59
Number analyzed (Eyes) | 122 | 118
logMAR
  2-Week Follow-up | -0.107 (0.0673) | -0.080 (0.0663)
  4-Week Follow-up | -0.106 (0.0713) | -0.091 (0.0678)
  8-Week Follow-up | -0.115 (0.0776) | -0.0881 (0.0665)
  12-Week Follow-up | -0.105 (0.0769) | -0.0892 (0.0686)

3. Primary Outcome: Percentage of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit lamp findings were graded using a FDA Grade Scale, 0 = None, 1 = Slight, 2 = Moderate, 3 = Significant, 4 = Advanced. Measurements were taken in each subject eye at the initial visit, 2-4-8- and 12-week follow-ups. A new response variable was derived by dichotomizing the data as follows: 1 if a Grade 3or higher SLF was observed and 0 otherwise. The Percentage of eyes with Grade 3 or higher SLFs was reported for each lens and time point.
Time Frame: Up to 12-Week Follow-up
Population: All subjects that were dispensed at least one study lens.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Senofilcon A With New UV Blocker (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 67 | 64
Number analyzed (Eyes) | 134 | 128
Percentage of eyes
  2-Week Follow-up | 0 | 0
  4-Week Follow-up | 0 | 0
  8-Week Follow-up | 0 | 0
  12-Week Follow-up | 0 | 0

4. Secondary Outcome: Contact Lens Wearing Time
Description: Contact lens wearing time (hours) was self-reported by each subject at the 2-, 4-, 8- and 12-week follow-ups. The average contact lens wearing time (hours) for each lens and time point was reported.
Time Frame: Up to 12-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Senofilcon A With New UV Blocker (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 61 | 59
Hours
  2-Week Follow-up | 14.7 (1.76) | 14.0 (2.14)
  4-Week Follow-up | 14.5 (2.03) | 14.2 (2.14)
  8-Week Follow-up | 14.6 (1.78) | 14.1 (2.02)
  12-Week Follow-up | 14.7 (1.67) | 14.3 (1.83)

5. Secondary Outcome: Percentage of Eyes With Subject Reported Symptoms Problems or Complaints
Description: Symptoms, problems and complaints are subject reported and were collected for each subject eye at the 1-, 2-, 4-, 8- and 12-week follow-up evaluations. The data is reported as a binary outcome of yes if a subject experience a problem or complaint or no otherwise. Symptoms, problems and complaints include the following: Burning/Stinging, Itchiness/Scratchiness, Dryness, Lens Awareness, Grittiness/Foreign Body Sensation, Redness, Irritation/Discomfort, Cloudy/Blurry/Hazy, Variable Vision and Other The Percentage of subjects eyes with symptoms, problems or complaints was reported for each lens and time point.
Time Frame: Up to 12-Week Follow-up
Population: All subjects that were dispensed at least one study lens.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Senofilcon A With New UV Blocker (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 67 | 64
Number analyzed (Eyes) | 134 | 128
Percentage of eyes
  1-Week Follow-up | 12.9 | 13.3
  2-Week Follow-up | 15.2 | 23.3
  4-Week Follow-up | 14.1 | 11.3
  8-Week Follow-up | 14.1 | 16.9
  12-Week Follow-up | 12.7 | 10.7

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of study lens wear. Approximately 12-weeks per subject.
Arm/Group | Senofilcon A With New UV Blocker | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/64
Other Adverse Events (participants affected / at risk) | 0/67 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02982018/SAP_000.pdf
  • Study Protocol (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02982018/Prot_001.pdf